CLINICAL TRIAL: NCT03360552
Title: Evaluating the Effectiveness of a New Way of Organizing Primary Health Care to Improve the Management of Alzheimer's Disease EvaMMADom
Brief Title: Evaluating the Effectiveness of a New Way of Organizing Primary Health Care to Improve the Management of Alzheimer's Disease
Acronym: EvaMMADom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-54; 2017-A01582-51 (Registry Identifier: IDRCB)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the multidimensional score of fragility (RAI CA) (Experimental): A general practitioner (MG) management strategy guided by a multidimensional evaluation (RAI-CA) on the multidimensional score of fragility (RAI-HC) of patients with mild to moderately severe dementia.
  Interventions: Other: Multidimensional fragility index questionnaire RAI-Home Care
- Usual care (Placebo Comparator): support for patients without multidimensional evaluation (RAI-CA)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Multidimensional fragility index questionnaire RAI-Home Care — Questionnaire for assessing deficits in Alzheimer's disease
  Arms: the multidimensional score of fragility (RAI CA)
Other: Usual care — Usual clinical evaluation
  Arms: Usual care

SUMMARY:
The objective of the present study is to evaluate the effectiveness of a general practitioner (MG) management strategy guided by a multidimensional evaluation on the multidimensional score of fragility of patients with mild to moderately severe dementia, compared to those currently implemented (without the provision of such an assessment). The measurement of the respective effectiveness of the two types of care in primary care will itself be based on a multidimensional evaluation performed independently in the memory center having established the diagnosis of Alzheimer's disease. The secondary objectives are the evaluation of the impact of the strategy on the functional abilities of patients, the incidence of geriatric syndromes, cognitive functions, quality of life of the patient and the burden of the primary caregiver. The efficiency of the strategy will be assessed through a cost-effectiveness analysis. A survey of opinions will also be conducted among primary health care providers, carers and CMs on the implemented system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with probable Alzheimer's disease, according to the criteria usually used in memory centers
* Aged over 64 years with mild to moderately severe dementia syndrome
* Volunteers for medical follow-up for a period of 20 months; Which the general practitioner attending agrees to participate in the research

Exclusion Criteria:

* Patients under 65 years old
* presenting with early cognitive decline or severe dementia
* Not meeting the clinical diagnostic criteria for Alzheimer's disease
* Refusing or unable to sign informed consent to participate
* Not voluntary for medical follow-up for a period of 20 months
* Whose general practitioner refuses to participate in the research

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of multidimensional fragility scores | 20 months
  The multidimensional evaluation score produced by Nurses in the home of AM patients and passed on to patients' doctors increases decision-making and patient care

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No